CLINICAL TRIAL: NCT03323203
Title: Association of Intraoperative Cerebral and Somatic Tissue Oxygen Saturation With Postoperative Acute Kidney Injury in Adult Patients Undergoing Double Valves Replacement Surgery
Brief Title: Association of Tissue Oxygen Saturation With Postoperative Acute Kidney Injury in Double Valves Replacement Surgery
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, chonglei, M.D.& Ph.D., Xijing Hospital
Other Study IDs: KY20172070-1
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FORE-SIGHT Elite, CASMED, Inc., Branford, Connecticut, USA — Tissue oxygenation was monitored using a tissue oximeter based on near-infrared spectroscopy (FORE-SIGHT Elite, CASMED, Inc., Branford, Connecticut, USA). The oximeter had four cables with each cable connected to an adhesive probe.

SUMMARY:
To investigate the relationship of tissue oxygenation of different organs and tissue beds (e.g., a tissue bed on the arm vs. leg vs. flank tissue bed(s) and renal tissue bed, and thus can be used as a surrogate of renal tissue oxygenation monitoring.

DETAILED DESCRIPTION:
In this study, we will monitor tissue oxygenation of four different tissue beds including cerebral tissue (SctO2) on the forehead, and 3 somatic tissue beds monitored on the forearm (SarmO2), upper leg (SlegO2), and the renal region (SrrO2). The primary end point is AKI and the secondary end points are postoperative major non-renal complications (e.g. stroke, delirium, myocardial infraction, heart failure, new or worsening arrhythmia, mechanical ventilation > 24 hours, deep wound infection, etc.) and mortality. The associations between tissue oxygenation of different tissue beds, i.e. SctO2, SarmO2, SlegO2, and SrrO2, and AKI and non-renal outcomes will be compared to explore the tissue bed(s) whose oxygen saturation has a stronger association with the outcomes of interest. The strength of this study is to use the patient as self-control.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Age ≥18 years of age
* Double valves replacement surgery with cardiopulmonary bypass (CPB)

Exclusion Criteria:

* The Trauma, deformity or abnormality sites which the sensor will be put may affect the monitoring of the data
* Preoperative renal dysfunction needs renal replacement therapy
* Emergency surgery
* Preoperative intubated patient
* Unable to cooperate with the study, i.e., mental illness, et al
* Patients with hemoglobin and anemia
* Participate in other trials in the prior 3 months
* Patient refuses to participate in the study
* Patient is unfit for the study decided by reach stuff

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to have double valves replacement surgery
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury (AKI) | Seven days postoperatively
  AKI is defined as any of the following (Not Graded):
  * K Increase in serum creatinine (SCr) by X0.3 mg/dl (X26.5 lmol/l) within 48 hours; or
  * K Increase in SCr to X1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  * K Urine volume o0.5 ml/kg/h for 6 hours.AKI is defined as any of the following (Not Graded):
  * K Increase in SCr by X0.3 mg/dl (X26.5 lmol/l) within 48 hours; or
  * K Increase in SCr to X1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  * K Urine volume o0.5 ml/kg/h for 6 hours.
  AKI is defined as any of the following (Not graded):Increase in SCr by X0.3 mg/dl (X26.5 lmol/l) within 48 hours; or increase in SCr to X1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or urine volume less than 0.5 ml/kg/h for 6 hours.

SECONDARY OUTCOMES:
Length of mechanical ventilation | Postoperative day 0-day 7
  Time between intubation and extubation
Length of ICU stay | Postoperative day 0-day 7
  Days between end of operation and departure of ICU
Length of hospital stay | Postoperative day 0-day 30
  Days between end of operation and hospital discharge
Adverse events in 30 days | Postoperative day 0-day 30
  Clinical events since hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Zhang T, Hou L, Zhao J, Fan Q, Wang L, Lu Z, Dong H, Lei C. Association of intraoperative cerebral and somatic tissue oxygen saturation with postoperative acute kidney injury in adult patients undergoing multiple valve surgery. BMC Anesthesiol. 2023 Sep 19;23(1):319. doi: 10.1186/s12871-023-02279-7. PMID 37726660